CLINICAL TRIAL: NCT06893198
Title: Conquering Hypertension in Urban Vietnam
Acronym: HTN-URBAN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Health Strategy and Policy Institute (Unknown)
Responsible Party: Principal Investigator, Hoa Nguyen, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H00001666; R61HL172269 (NIH)
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
Keywords: storytelling intervention; home blood pressure monitoring; community health workers; Urban hypertension; Vietnam; HTN-URBAN intervention
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison Group (Active Comparator): Patients in the comparison group will receive the "Learn More" module only.
  Interventions: Behavioral: "Learn More" module only
- Intervention Group (Experimental): Patients in the intervention group will receive HTN-URBAN intervention, which includes three integrated components:
  (1) Storytelling intervention, (2) Home BP monitoring, (3) Expanded community health worker services.
  Interventions: Behavioral: Storytelling intervention; Behavioral: Home BP monitoring; Behavioral: Expanded community health worker services

INTERVENTIONS:
Behavioral: Storytelling intervention — The storytelling intervention consists of interactive, literacy-appropriate, and culturally sensitive multimedia storytelling modules for motivating behavior change through the power of patients speaking in their own voice. Based on preferences that emerged during the researchers' formative work with the partnering rural communities, the storytelling intervention will be delivered via Computerized Intervention Authoring System (CIAS) on a biweekly basis. A supplementary "Learn More" module of didactic material (3 minutes) provides strategies for better patient-physician communication and is coordinated with the specific patient stories will be provided via CIAS as well.
  Arms: Intervention Group
Behavioral: Home BP monitoring — Patients with hypertension will be provided blood pressure monitors and guided to self-measure their blood pressure and to record their blood pressure daily at home.
  Arms: Intervention Group
Behavioral: Expanded community health worker services — A training program will be implemented for community health workers for the intervention arm regarding hypertension management at the community level so that they can assist patients better managing their blood pressure at home.
  Arms: Intervention Group
Behavioral: "Learn More" module only — A supplementary "Learn More" module of didactic material (3 minutes) provides strategies for better patient-physician communication, which will be delivered via Computerized Intervention Authoring System (CIAS) at baseline and at 3, 6, and 9 months after enrollment.
  Arms: Comparison Group

SUMMARY:
The HTN-URBAN project aims to improve hypertension (HTN) control for adults in a large northern Vietnamese city via a cluster-randomized trial design.

DETAILED DESCRIPTION:
A Cluster-randomized, Type II Hybrid effectiveness implementation Trial will take place in 14 urban communities in 7 urban districts in Hai Phong city in northern Vietnam.

Community Eligibility Criteria: (1) located in urban Hai Phong city; (2) distance between 2 communities will be at least 10 Km; (3) no other research studies/ health programs currently being implemented; and (4) key community and clinical leaders are willing to participate in the study.

Recruitment

Residents from participating sites will be invited to attend the community screening events run by local community health center (CHC) staff and Community Health Workers (CHWs). Those meeting our pre-defined eligibility criteria will be invited to their CHCs to learn more about the study. Patients with elevated blood pressure (BP) will be invited for re-measurement over the next two weeks (at least 1 week apart). After the second BP measurement, patients with elevated BP will be invited to participate in the study.

Randomization

Fourteen communities in urban Hai Phong (700 patients with uncontrolled hypertension - HTN) will be randomly assigned either to an intervention (7 communities- 50 patients per community) or comparison group (7 communities- 50 patients per community) by a computer procedure. Patients with uncontrolled HTN will be assigned to intervention versus comparison status based on the communities in which they reside.

Intervention group: The intervention group will receive 3 components including digital Storytelling delivered via Computerized Intervention Authoring System (CIAS), home blood pressure self-monitoring and expanded CHW services (frequent contacts, visits and consultations).

Comparison group: Patients in the comparison group will receive only "Learn More" module - didactic material without HTN related stories via CIAS.

Patients in both groups will be followed up at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old;
* Presence of uncontrolled HTN (systolic BP ≥ 140 mmHg or diastolic BP ≥ 90 mmHg) according to JNC-8;
* Willing to provide informed consent.

Exclusion Criteria:

* Participation in another study on hypertension;
* Pregnant;
* Advanced cognitive impairment;
* Previous exposure to storytelling modules;
* Participant family member;
* Participant in intervention development.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure level | From baseline to 3, 6 and 12 month follow up visits
  Changes in systolic blood pressure levels
Acceptability, Appropriateness, Feasibility | at 3, 6, and 12 month follow-up visits
  Information will be collected via semi-structured interviews among patients, Community health workers, community leaders, and local clinicians and nurses mentioned previously and patient interviews and post-story viewing surveys.
Adoption | at baseline, 3, 6, and 12 month follow-up visits
  Data for participant recruitment and retention will include the number of patients approached for recruitment, reasons for ineligibility of patients not enrolled or refusing to participate, and completion rates for follow-up visits.
Fidelity | at 3, 6, and 12 month follow-up visits
  Information will be collected via periodic random observations of blood pressure measurement and patient interviews by study investigators and the project manager who will document and check intervention deliverables using a standardized checklist.

SECONDARY OUTCOMES:
Diastolic blood pressure level | From baseline to 3, 6 and 12 months
  Changes in diastolic blood pressure levels
Hypertension control | From 3 to 6 and12 months follow up visits
  Changes in the proportion of patients with hypertension control.
Self-efficacy | From baseline to follow-up at 3, 6, and 12 months
  Changes in patients medication adherence self-efficacy, which will be measured using the Medication Adherence Self-efficacy Scale (MASES) instrument.
Hypertension (HTN) medication adherance | From baseline to 3, 6, and 12 month follow-up visits
  Changes in adherence to anti-HTN medications, which will be measured using a standardized data collection form.
Risk of cardiovascular disease (CVD) | From baseline to follow-up at 12 months
  Changes in CVD risk factors (tobacco use, alcohol consumption, salt intake and physical activities), which will be measured using WHO STEPs questionnaires
Patient quality of life | From baseline to 3, 6 and 12 month follow up visits
  Changes in patient's quality of life, which will be measured using the SF-12 survey.
Cost | at 12 month follow up
  Program costs and patient-related costs will be collected.
  Program costs include intervention development and its implementation at the district and community levels: personnel, equipment, medical devices, training materials and supplies, transportation, administration, and other operational expenses.
  Patient-related costs include medications, time lost from work, Community Health Center visits, and consultation fees and patient utilities will be collected using a survey administered at the final visit.

CONTACTS AND LOCATIONS:
Overall Officials: Hoa Nguyen, MD, MS, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- Health Strategy and Policy Institute, Hanoi, Vietnam, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data that will be collected for this study can be obtained by contacting the study PI.
Supporting Information: Study Protocol, SAP
Time Frame: The final dataset will be available from January 2030 to December 2039.
Access Criteria: The data and associated documentation will be available to qualified academic investigators for non-commercial research under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Ha DA, Tran OT, Nguyen HL, Chiriboga G, Goldberg RJ, Phan VH, Nguyen CT, Nguyen GH, Pham HV, Nguyen TT, Le TT, Allison JJ. Conquering hypertension in Vietnam-solutions at grassroots level: study protocol of a cluster randomized controlled trial. Trials. 2020 Nov 27;21(1):985. doi: 10.1186/s13063-020-04917-8. PMID 33246495
- [Background] Nguyen HL, Ha DA, Goldberg RJ, Kiefe CI, Chiriboga G, Ly HN, Nguyen CK, Phan NT, Vu NC, Nguyen QP, Allison JJ. Culturally adaptive storytelling intervention versus didactic intervention to improve hypertension control in Vietnam- 12 month follow up results: A cluster randomized controlled feasibility trial. PLoS One. 2018 Dec 31;13(12):e0209912. doi: 10.1371/journal.pone.0209912. eCollection 2018. PMID 30596749
- [Background] Allison JJ, Nguyen HL, Ha DA, Chiriboga G, Ly HN, Tran HT, Phan NT, Vu NC, Kim M, Goldberg RJ. Culturally adaptive storytelling method to improve hypertension control in Vietnam - "We talk about our hypertension": study protocol for a feasibility cluster-randomized controlled trial. Trials. 2016 Jan 14;17:26. doi: 10.1186/s13063-015-1147-6. PMID 26762128
- [Background] Ha DA, Tran OM, Nguyen HL, Nguyen HT, Dao AM, Nguyen HV, Vu NC, Chiriboga G, Goldberg RJ, Houston TK, Allison JJ. Stakeholder Engagement in Late-Stage Translation Phase 4 Research for Noncommunicable Diseases in Low- and Middle-Income Countries: What Works and Why-The Vietnam Experience (UMMS-Vietnam Team). Glob Heart. 2019 Jun;14(2):143-147. doi: 10.1016/j.gheart.2019.05.003. PMID 31324368
- [Background] Nguyen HL, Ha DA, Tran OT, Phan VH, Nguyen CT, Nguyen GH, Nguyen TT, Le TT, Goldberg RJ, Wang B, Tang ET, Chiriboga G, Budhwani H, Allison JJ. Conquering hypertension in Vietnam: 12- month follow up results from a cluster-randomised controlled trial. Lancet Reg Health West Pac. 2024 Jul 1;48:101123. doi: 10.1016/j.lanwpc.2024.101123. eCollection 2024 Jul. PMID 39045484